CLINICAL TRIAL: NCT06147115
Title: The Validation of Rockall Scoring System in Predicting Outcomes From Variceal Bleeding in Sudanese Patients: Cross-sectional Study.
Brief Title: The Validation of Rockall Scoring System in Predicting Outcomes From Variceal Bleeding
Status: Completed | Type: Observational
Sponsor: National Center for Gastroentestinal and Liver Disease (Other)
Responsible Party: Sponsor
Other Study IDs: GastroentestinalLiverRockall
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Bleeding Esophageal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment tool to determine severity of GI bleeding — The Rockall score is a validated mortality risk assessment for patients admitted with upper GI bleeding.

SUMMARY:
Objective This study aims to evaluate the validation of the Rockall scoring system in predicting the outcomes of variceal bleeding among Sudanese patients.

Design/Method A cross-sectional hospital-based study involved 150 adult Sudanese patients presenting with upper gastrointestinal bleeding (UGIB) of variceal origin. Patients with UGIB resulting from causes other than varices and those who declined participation were excluded. Data were collected through a structured questionnaire complemented by upper gastrointestinal tract endoscopy findings, and patients were followed up until discharge.

Results The study encompassed 150 patients, predominantly male (117, 78%), aged between 18 and 60 years (n=119, 79%), residing mainly in central regions (134, 89%). The leading presenting complaints included hematemesis (70, 46.7%) and melena (22, 14.6%). Notably, peri-portal fibrosis (101, 67.3%) and cirrhosis (24, 16%) were the primary etiological factors, with a significant prevalence of alcohol consumption (87, 58%). Concerning the grade of esophageal varices, grades III and IV were most prevalent (67, 44.7% and 47, 31.3%, respectively), and fundal varices were identified in 13 patients (8.7%). The mean Rockall score was 3.83 ± 1.99, indicating moderate severity. Additionally, the Rockall score showed significant associations with the number of sessions, complications, bleeding recurrence, duration of hospital stay, and mortality (p < 0.05).

Conclusion Understanding the significance of the Rockall scoring system and its applicability to Sudanese patients with variceal bleeding has the potential to guide more effective strategies in the management of upper gastrointestinal tract bleeding, ultimately improving patient outcomes and reducing morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older
* primary complaints of upper GI bleeding

Exclusion Criteria:

* Patients with upper GI bleeding resulting from causes other than varices
* who declined to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 patients were enrolled in the study between June and September 2012. The study comprised patients aged 18 years and older, presenting with upper gastrointestinal (GI) bleeding of variceal origin, who visited the outpatient and referral clinic at the center and reported primary complaints of upper GI bleeding (UGIB), including hematemesis and/or melena. Patients with upper GI bleeding resulting from causes other than varices, as well as those who declined to participate in the study, were excluded
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2012-09-10 (Actual)

PRIMARY OUTCOMES:
the validation of the Rockall scoring system in predicting the outcomes of variceal bleeding among Sudanese patients | June 2012 - Sep 2012
  The primary outcome measure in this study appears to be the validation of the Rockall scoring system in predicting the outcomes of variceal bleeding among Sudanese patients presenting to the Mohammed Salih Idris Bleeding Center (MSIBC). The study aims to assess the effectiveness of the Rockall scoring system in predicting mortality, bleeding recurrence, and other clinical outcomes in Sudanese patients with variceal bleeding. The Rockall scoring system incorporates various factors, including age, evidence of shock, coexisting medical conditions, and the presence of visible signs of hemorrhage. The study investigates the association between Rockall scores and clinical outcomes such as mortality, bleeding recurrence, complications, duration of hospital stay, and interventions conducted. The validation of the Rockall scoring system in the context of variceal bleeding in Sudan is crucial for risk stratification and guiding the management of patients with variceal bleeding.